CLINICAL TRIAL: NCT02382380
Title: Evaluation of Gadoterate in Patients With Renal Dysfunction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated by the Institutional Review Board
Sponsor: Loyola University (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 206338
Record Dates: First submitted 2015-02-27; First posted 2015-03-06 (Estimated); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Renal Dysfunction
Keywords: Magnetic Resonance Imaging; Contrast Agent; Gadoterate
MeSH Terms: conditions — Renal Insufficiency | interventions — gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gadoterate (Experimental): Patients who choose to receive Gadoterate will receive an MRI exam with standard pre-contrast and Gadoterate-enhanced acquisitions (0.2 mL/kg). The MRI protocol utilized in the study will be comprised of the standard Body protocols (routine abdomen, liver-pancreas, renal, prostate, angiography) as well as the standard Neurologic exam protocols (routine brain, orbital, brainstem, neck, angiography).
  Interventions: Drug: Gadoterate
- No Gadoterate (Other): Patients who choose not to receive Gadoterate will receive an MRI exam with no Gadolinium contrast. MRI protocols utilized in the study will be comprised of the standard Body protocols (routine abdomen, liver-pancreas, renal, prostate, angiography) as well as the standard Neurologic exam protocols (routine brain, orbital, brainstem, neck, angiography).
  Interventions: Other: No Gadoterate

INTERVENTIONS:
Drug: Gadoterate — Patients who choose to receive Gadoterate will receive an MRI exam with standard pre-contrast and Gadoterate-enhanced acquisitions (0.2 mL/kg). The MRI protocol utilized in the study will be comprised of the standard Body protocols (routine abdomen, liver-pancreas, renal, prostate, angiography) as well as the standard Neurologic exam protocols (routine brain, orbital, brainstem, neck, angiography).
  Other Names: Dotarem
  Arms: Gadoterate
Other: No Gadoterate — Patients who choose not to receive Gadoterate will receive an MRI exam with no Gadolinium contrast. The MRI protocol utilized in the study will be comprised of the standard Body protocols (routine abdomen, liver-pancreas, renal, prostate, angiography) as well as the standard Neurologic exam protocols (routine brain, orbital, brainstem, neck, angiography).
  Arms: No Gadoterate

SUMMARY:
This study is for individuals with decreased kidney function whose doctor has ordered Magnetic Resonance Imaging (MRI). Because kidney function is decreased, these patients usually do not receive the intravenous contrast material that can improve the accuracy of the MRI findings. The purpose of this study is to evaluate the safety and benefit of using a contrast material called Gadoterate in patients with decreased kidney function.

DETAILED DESCRIPTION:
Gadolinium-based intravenous contrast agents are widely used for the enhancement of MRI findings. However, these agents have been implicated in varying degrees of nephrotoxicity and therefore are not usually used in patients with renal dysfunction. Gadoterate is a Gadolinium agent and previous studies have indicated that it is safe in patients with decreased kidney function. The purpose of this study is to evaluate the safety and efficacy of using Gadoterate in this patient population.

Participants who have been scheduled for an MRI will choose to either receive Gadoterate contrast as part of their MRI or not receive Gadoterate as part of their MRI.

ELIGIBILITY:
Inclusion Criteria:

* Glomerular filtration rates (GFR) less than 30 ml/min but not on dialysis
* Being sent for an MRI examination in the course of routine clinical evaluation of one of the following indications: suspected or known head/neck/brain mass, hepatic mass, renal mass, pancreatic mass, or prostate mass, as well as evaluation of carotid or abdominopelvic vasculature.

Exclusion Criteria:

* Pregnant and lactating females
* Planned initiation of chemotherapy or surgery within 72 hours of the MRI exam
* Hemodynamic instability or acute coronary syndrome
* History of nephrotoxic medication within 2 weeks of the exam
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Goldberg, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomsen HS. Nephrogenic systemic fibrosis: A serious late adverse reaction to gadodiamide. Eur Radiol. 2006 Dec;16(12):2619-21. doi: 10.1007/s00330-006-0495-8. Epub 2006 Oct 24. No abstract available. PMID 17061066
- [Background] Sam AD 2nd, Morasch MD, Collins J, Song G, Chen R, Pereles FS. Safety of gadolinium contrast angiography in patients with chronic renal insufficiency. J Vasc Surg. 2003 Aug;38(2):313-8. doi: 10.1016/s0741-5214(03)00315-x. PMID 12891113
- [Background] Perazella MA. Current status of gadolinium toxicity in patients with kidney disease. Clin J Am Soc Nephrol. 2009 Feb;4(2):461-9. doi: 10.2215/CJN.06011108. PMID 19201920
- [Background] Janus N, Launay-Vacher V, Karie S, Clement O, Ledneva E, Frances C, Choukroun G, Deray G. Prevalence of nephrogenic systemic fibrosis in renal insufficiency patients: results of the FINEST study. Eur J Radiol. 2010 Feb;73(2):357-9. doi: 10.1016/j.ejrad.2008.11.021. Epub 2009 Jan 6. PMID 19128909
- [Background] Port M, Idee JM, Medina C, Robic C, Sabatou M, Corot C. Efficiency, thermodynamic and kinetic stability of marketed gadolinium chelates and their possible clinical consequences: a critical review. Biometals. 2008 Aug;21(4):469-90. doi: 10.1007/s10534-008-9135-x. Epub 2008 Mar 15. PMID 18344005
- [Background] Laurent S, Elst LV, Muller RN. Comparative study of the physicochemical properties of six clinical low molecular weight gadolinium contrast agents. Contrast Media Mol Imaging. 2006 May-Jun;1(3):128-37. doi: 10.1002/cmmi.100. PMID 17193689
- [Background] Deray G, Rouviere O, Bacigalupo L, Maes B, Hannedouche T, Vrtovsnik F, Rigothier C, Billiouw JM, Campioni P, Ferreiros J, Devos D, Alison D, Glowacki F, Boffa JJ, Marti-Bonmati L. Safety of meglumine gadoterate (Gd-DOTA)-enhanced MRI compared to unenhanced MRI in patients with chronic kidney disease (RESCUE study). Eur Radiol. 2013 May;23(5):1250-9. doi: 10.1007/s00330-012-2705-x. Epub 2012 Dec 5. PMID 23212275
- [Background] Maurer M, Heine O, Wolf M, Durmus T, Wagner M, Hamm B. Tolerability and diagnostic value of gadoteric acid in the general population and in patients with risk factors: results in more than 84,000 patients. Eur J Radiol. 2012 May;81(5):885-90. doi: 10.1016/j.ejrad.2011.04.022. Epub 2011 May 8. PMID 21555197
- [Background] Herborn CU, Honold E, Wolf M, Kemper J, Kinner S, Adam G, Barkhausen J. Clinical safety and diagnostic value of the gadolinium chelate gadoterate meglumine (Gd-DOTA). Invest Radiol. 2007 Jan;42(1):58-62. doi: 10.1097/01.rli.0000248893.01067.e5. PMID 17213750
- [Background] Broome DR, Girguis MS, Baron PW, Cottrell AC, Kjellin I, Kirk GA. Gadodiamide-associated nephrogenic systemic fibrosis: why radiologists should be concerned. AJR Am J Roentgenol. 2007 Feb;188(2):586-92. doi: 10.2214/ajr.06.1094. PMID 17242272
- [Background] Lencioni R, de Baere T, Burrel M, Caridi JG, Lammer J, Malagari K, Martin RC, O'Grady E, Real MI, Vogl TJ, Watkinson A, Geschwind JF. Transcatheter treatment of hepatocellular carcinoma with Doxorubicin-loaded DC Bead (DEBDOX): technical recommendations. Cardiovasc Intervent Radiol. 2012 Oct;35(5):980-5. doi: 10.1007/s00270-011-0287-7. Epub 2011 Oct 19. PMID 22009576
- [Background] Lima XT, Alora-Palli MB, Kimball AB, Kay J. Validation of a screening instrument for nephrogenic systemic fibrosis. Arthritis Care Res (Hoboken). 2013 Apr;65(4):637-42. doi: 10.1002/acr.21877. PMID 23097320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on November 5, 2014 and ended on May 15, 2019
Period: Overall Study
Arm/Group | Gadoterate | No Gadoterate
Started | 33 | 13
Completed | 31 | 10
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Gadoterate | Gadoterate | Total
Number analyzed (Participants) | 13 | 33 | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57.2 [49.0 to 63.1] | 64.2 [52.3 to 71.2] | 59.5 [49.1 to 68.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 16 | 21
  Male | 8 | 17 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 12 | 28 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 7 | 23 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 33 | 46
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 30.5 [29.8 to 36.3] | 28.6 [26.3 to 31.3] | 29.6 [26.3 to 31.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: Change in GFR from 0 to 72 hours
Time Frame: 72 hours
Population: The analysis population includes all participants with a baseline and 72-hour follow-up GFR assessment
Measure: Median (Inter-Quartile Range); unit: ml/minute
Arm/Group | No Gadoterate | Gadoterate
Number analyzed (Participants) | 10 | 31
ml/minute | 1.5 [1.0 to 5.0] | 1.0 [-2.0 to 3.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 3 years
Arm/Group | No Gadoterate | Gadoterate
All-Cause Mortality (participants affected / at risk) | 0/13 | 5/33
Serious Adverse Events (participants affected / at risk) | 0/13 | 5/33
Other Adverse Events (participants affected / at risk) | 0/13 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Gadoterate (N=13) | Gadoterate (N=33)
Cancer exacerbation leading to death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02382380/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02382380/ICF_001.pdf